CLINICAL TRIAL: NCT01794546
Title: Integrated Care for Pediatric Obesity Using Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Cara Ebbeling, Associate Director, New Balance Foundation Obesity Prevention Center, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5781
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Pediatric Obesity
Keywords: pediatric obesity; telehealth
MeSH Terms: conditions — Pediatric Obesity | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Telehealth (Experimental): The "immediate" intervention group will receive the telehealth intervention during the first 6 months of the study timeline.
  Interventions: Behavioral: Telehealth
- Wait List Control (Active Comparator): The "wait list" control group will receive the telehealth intervention during months 6 through 12 of the study timeline.
  Interventions: Behavioral: Telehealth

INTERVENTIONS:
Behavioral: Telehealth — Telehealth visits will alternate between a dietitian and behavioral medicine provider for either 30 minutes or 1 hour. Over a 6-month period, 12 telehealth sessions will be scheduled for each participant. The dietitian will provide dietary and physical activity recommendations, and the behavioral medicine provider will counsel on strategies for achieving specific goals. Applying a Chronic Care Model, self-management support will be augmented by linkages to community resources.

SUMMARY:
Obesity is perhaps the most urgent public health crisis in pediatrics. Thus, managing childhood obesity is a top priority among pediatricians in primary care settings. However, effective treatment typically is multidisciplinary, and most practices currently do not have the infrastructure for coordinating integrated care. With the advent of the Affordable Care Act (ACA), innovative systems for building multidisciplinary teams to provide integrated care through a patient-centered medical home will be at a strategic advantage. The use of electronic technologies for delivering health-related information or services, known as telehealth, is an innovation with the potential to streamline integrated care and transform interventions for chronic diseases. We propose a pilot study to evaluate telehealth for treating pediatric obesity in collaboration with a community practice (Wareham Pediatrics).

Patients aged 10 to 17 years who participate in the telehealth intervention study (N=40) will be randomly assigned to an "immediate" intervention group or a "wait list" control group. Subjects in the "immediate" intervention group will begin the 6-month telehealth intervention at the time of enrollment in the study and then receive general patient/family counseling from their primary care providers (PCPs) at routine office visits during a 6-month follow-up period. Those in the "wait list" control group will receive general patient/family counseling from their PCPs for 6 months followed by the telehealth intervention for 6 months. Thus, the total duration of participation in the study for each subject will be 12 months. The telehealth intervention will include dietary, physical activity, and behavioral management counseling provided by videoconferencing from the OWL clinical providers at Boston Children's Hospital to children in their homes, or at a telehealth station at Wareham Pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 17 years
* BMI ≥95th percentile for age and sex
* No known significant obesity comorbidity or cause requiring urgent medical evaluation or treatment in a subspecialty program other than an obesity program
* No known physical limitations to changes in diet or activity level (i.e., concern for cardiac disease, primary gastrointestinal disease, or orthopedic concerns)
* Patient at Wareham Pediatrics practice

Exclusion Criteria:

* Unstable home environment (homeless, temporary living situation, lack of working phone or electricity)
* Inability to actively participate in treatment (developmental delay, nonverbal, severe psychiatric illness).
* Physician diagnosis of a major medical illness or eating disorder.
* Chronic use of any medication or supplement that may affect study outcomes.
* Another member of the family (i.e., first degree relative) or household participating in the study.
* Planning to relocate from current area of residence during the proposed timeframe for study participation

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
BMI | 12 months
  Hypotheses. 1) The mean decrease in body mass index (BMI) percentile at 6 months (primary outcome) will be greater among subjects who are randomly assigned to the "immediate" intervention group compared to the "wait list" control group. 2) For children in the "immediate" intervention group, the intervention effect on BMI percentile will be maintained during a 6-month follow-up period. 3) For children in the "wait list" control group, BMI percentile will improve during the 6-month delayed telehealth intervention period compared to the initial 6-month control period.

SECONDARY OUTCOMES:
Satisfaction and compliance | 12 months
  Hypotheses. 1) Satisfaction with the intervention will be higher at 6 months for the "immediate" intervention group vs. "wait list" control group. 2) Subjects in both groups (during either the "immediate" or "delayed" telehealth intervention, depending on random assignment) will complete a higher percentage of scheduled telehealth intervention visits (≥75%) when compared to published data of completed in-person visits from a national survey of established weight management clinics in children's hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Cara B. Ebbeling, PhD, Principal Investigator — Boston Children's Hospital; Amy D Fleischman, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Wareham Pediatrics, Wareham, Massachusetts, United States

REFERENCES:
- [Background] Ebbeling CB, Feldman HA, Chomitz VR, Antonelli TA, Gortmaker SL, Osganian SK, Ludwig DS. A randomized trial of sugar-sweetened beverages and adolescent body weight. N Engl J Med. 2012 Oct 11;367(15):1407-16. doi: 10.1056/NEJMoa1203388. Epub 2012 Sep 21. PMID 22998339
- [Background] Ebbeling CB, Leidig MM, Feldman HA, Lovesky MM, Ludwig DS. Effects of a low-glycemic load vs low-fat diet in obese young adults: a randomized trial. JAMA. 2007 May 16;297(19):2092-102. doi: 10.1001/jama.297.19.2092. PMID 17507345
- [Background] Ebbeling CB, Leidig MM, Sinclair KB, Hangen JP, Ludwig DS. A reduced-glycemic load diet in the treatment of adolescent obesity. Arch Pediatr Adolesc Med. 2003 Aug;157(8):773-9. doi: 10.1001/archpedi.157.8.773. PMID 12912783
- [Background] Fleischman A, Kron M, Systrom DM, Hrovat M, Grinspoon SK. Mitochondrial function and insulin resistance in overweight and normal-weight children. J Clin Endocrinol Metab. 2009 Dec;94(12):4923-30. doi: 10.1210/jc.2009-1590. Epub 2009 Oct 21. PMID 19846731
- [Background] Fleischman A, Makimura H, Stanley TL, McCarthy MA, Kron M, Sun N, Chuzi S, Hrovat MI, Systrom DM, Grinspoon SK. Skeletal muscle phosphocreatine recovery after submaximal exercise in children and young and middle-aged adults. J Clin Endocrinol Metab. 2010 Sep;95(9):E69-74. doi: 10.1210/jc.2010-0527. Epub 2010 Jun 16. PMID 20554709
- [Background] McCormack SE, McCarthy MA, Farilla L, Hrovat MI, Systrom DM, Grinspoon SK, Fleischman A. Skeletal muscle mitochondrial function is associated with longitudinal growth velocity in children and adolescents. J Clin Endocrinol Metab. 2011 Oct;96(10):E1612-8. doi: 10.1210/jc.2011-1218. Epub 2011 Aug 10. PMID 21832105
- See also: Related Info — http://www.warehampeds.com/